CLINICAL TRIAL: NCT06103006
Title: Remote Physiotherapy to Protect Physical Health in Duchenne Muscular Dystrophy: Telerehabilitation
Brief Title: Remote Physiotherapy to Protect Physical Health in Duchenne Muscular Dystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Mustafa Sarı, Research Assistant, Lokman Hekim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 003/2021
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation Group (Experimental): Participants in this group will receive telerehabilitation exercises.
  Interventions: Other: Telerehabilitation

INTERVENTIONS:
Other: Telerehabilitation — The structured telerehabilitation program focused on 4 specific objectives: breathing, stretching, posture, and stability. The duration was between 20-30 minutes. Exercises involving the major muscle groups (upper, lower extremity, and trunk muscle groups) were applied by the physiotherapists. Strengthening and stretching sets and repetitions were started with 1 set of 8-15 reps (progress to >1 set).

SUMMARY:
Duchenne Muscular Dystrophy (DMD) is a progressive genetic neuromuscular disease characterized by progressive loss of motor function, respiratory failure, and cardiomyopathy required regular physiotherapy. With the outbreak of the pandemic rehabilitation centers that make up the weekly physiotherapy routine of children with disabilities have slowed down or even stopped their activities. So DMD who have additional diseases such as respiratory muscle weakness, spinal deformity, obesity, and cardiac dysfunction have also been negatively affected. The 'telerehabilitation' method, which is well planned and prepared for the abilities and needs of patients and caregivers, is seen as a good option at this point.

Studies, reporting the feasibility and safety of telerehabilitation in joint replacement, multiple sclerosis, and post-operative conditions, report that the length of stay was reduced, there was access to the same level of service regardless of the distance, and there was no travel cost. Despite these advantages, the framework and applicability of telerehabilitation programs have been investigated limited and not focused on effectiveness of telerehabilitation in patients with DMD.

According to the current knowledge, telerehabilitation in DMD is a subject that needs to be investigated in terms of its benefits. So, in this study, it was aimed to show the telerehabilitation's feasibility and its effects on performance level, endurance, fall frequency, pulmonary functions, and satisfaction level with the program in individuals with DMD.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate verbally and visually,
* Older than 5 years old

Exclusion Criteria:

* Individuals who had undergone any surgical operations in the past 6 months,
* Had a severe cognitive and breathing impairment,
* Using mechanical ventilator continually or intermittent,
* Having febrile infection

Ages: 5 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Endurance | Change from baseline at 8 weeks
  Number of times the individuals can flexed and extend their knees in a sitting position for 30 seconds. Also, the number of elbow flexion/extension was recorded
Modified Upper Extremity Performance Test | Change from baseline at 8 weeks
  Flexion the shoulder to 90 degrees, flexion the shoulder above 90 degrees (above eye level), abduction of the shoulder 90 degrees, abduction of the shoulder above 90 degrees, doing the same movements with weight, bringing the empty glass to the mouth in a sitting position, bringing the full glass to the mouth were evaluated. It was scored as 0 point (cannot), 1 point (can do with compensation), 2 points (does independently). In addition, the time to pick up 5 coins (50 cents size coin or similar) on the table with one hand was recorded .

SECONDARY OUTCOMES:
10 Meter (m) Walking Test | Change from baseline at 8 weeks
  The distance of 10 m was determined in a suitable indoor environment, the individual was asked to walk this distance and the time that the patient walked was recorded.
Stand Up from the Supine Position Test | Change from baseline at 8 weeks
  Depending on the severity of the disease, this period is extended. Depending on the weakness of the hip and shoulder girdle and trunk muscles, there is a movement model that the individuals use by climbing over himself. While the individual is getting up from the ground, the mother and the physiotherapist keep time with a stopwatch.
Single Breath Count (SBC) | Change from baseline at 8 weeks
  Single breath count (SBC) is the maximum measure of serial counting of numbers in normal speaking voice after a maximal inhalation. SBC has good correlation with the gold standard measures of pulmonary function test (PFT), peak expiratory flow rate (PEFR), and forced expiratory volume in the first second (FEV1). The value reached is recorded when the patient counts audibly in a single expiration after maximum inspiratory effort. The instruction is: "Breathe well, count as many counts as possible while exhaling". The total number is recorded and evaluated in 4 categories: >30: 1, 20-29:2, 10-19: 3, <9:4.
Patient Satisfaction Survey | After 8 weeks
  15 items survey was developed by the researchers. 5 likert pointed scale range was "5: excellent" and "1=bad". The items were about internet/connection, physiotherapist's guidance, timing, level of knowledge, reassurance, comfort, information/suggestions, the intelligibility of information, and general satisfaction. A total score was used to calculate percent value [(100 X Total score)/15].
Brooke Upper Extremity Scale | Change from baseline at 8 weeks
  The Brooke scale was used to classify upper extremity functioning with scores from 1 to 6 (higher scores indicate worse functionality).
Brooke Lower Extremity Scale | Change from baseline at 8 weeks
  The functional ability for all of the subjects with DMD was also ranked by a physical therapist using the Brooke Lower Extremity Functional Scale. This scale ranges from a grade of 1 (able to walk and climb stairs independently) to a grade of 10 (confined to bed).
Frequency of falling | Change from baseline at 8 weeks
  The number of falls that occurred per day before the study and the frequency of falls after 8 weeks of exercise were questioned verbally.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Turkey (Türkiye)